CLINICAL TRIAL: NCT02763644
Title: A Randomized, Open Label, Controlled, Multiple Dose Study to Evaluate the Clinical Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LFG316 in Patients With Transplant Associated Microangiopathy After Hematopoietic Precursor Cell Transplantation
Brief Title: Efficacy and Safety of LFG316 in Transplant Associated Microangiopathy (TAM) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: LFG316, had been studied in seven patients with transplantation-associated microangiopathy. Due to low confidence of clinical benefit, this study was closed.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLFG316X2202
Record Dates: First submitted 2016-04-14; First posted 2016-05-05 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Transplant Associated Microangiopathy TAM
Keywords: transplant associated microangiopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LFG316 plus SoC (Experimental): LFG316 plus SoC (excluding plasmapheresis and prohibited treatment)
  Interventions: Drug: LFG316 active drug; Other: Standard of care treatment
- All SoC first (Experimental): Standard of Care then LFG316 plus SoC
  Interventions: Drug: LFG316 active drug; Other: Standard of care treatment

INTERVENTIONS:
Drug: LFG316 active drug — LFG316
  Other Names: LFG316
Other: Standard of care treatment — SoC (site specific)
  Other Names: SoC

SUMMARY:
This was a randomized, SoC-controlled, open-label, multi-center study in patients with TAM after hematopoietic precursor cell transplantation (HPCT) .

Study consisted of up to 28 days of screening period, 16 weeks treatment period that can be extended to 45 weeks.Approximately 40 patients was to be randomized to receive SoC or LFG316 plus SoC. Patients was included in the study if they have diagnosis of TAM and poor prognostic markers. This trial was terminated: LFG316, a monoclonal antibody inhibitor of complement factor 5 (C5), had been studied in seven patients with transplantation-associated microangiopathy (TAM). Due to low confidence of clinical benefit, this study was closed

DETAILED DESCRIPTION:
This was a randomized, SoC-controlled, open-label, multi-center study in patients with TAM after hematopoietic precursor cell transplantation (HPCT). Study consisted of up to 28 days of screening period, 16 weeks treatment period that can be extended to 45 weeks, 36 weeks follow up, and end of study visit (EOS) at week 52. Duration of follow up depended on duration of treatment. Patients who are treated for more than 41 weeks will proceed directly to EOS visit.

Approximately 40 patients was to be randomized to receive SoC or LFG316 plus SoC. Patients was included in the study if they have diagnosis of TAM and poor prognostic markers.

Patients showing worsening of disease after two weeks of treatment or showing no response at week 4 or any time after will be considered failures and can be switched to receive the alternative treatment (SoC or LFG316). Patients can only switch treatment arms once.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent before any study-specific screening procedures. For pediatric patients, consent will be obtained from parent(s) or legal guardian(s) and the signature of at least 1 parent or guardian will be required. Investigators will also obtain assent of patients according to local, regional or national guidelines.
2. Patients after allogeneic stem cell transplantation from a related or unrelated, HLA-matched or mismatched donor with the diagnosis of transplant related microangiopathy. Patients having received any of the following stem cell sources are eligible: G-CSF mobilized peripheral blood stem cells, bone marrow, umbilical cord blood.
3. Male and female TAM patients ≥ 2 years old at the time of first dose administration. Patients < 12 years old can only be included in the study after first IA has shown that it is safe and well tolerated in patients ≥ 12 years old (Section 3.5).
4. The presence of TAM as per below diagnostic criteria at baseline (or screening if baseline visit is skipped). All the criteria have to be met for the patients included in the study:

   * Elevated lactate dehydrogenase (any elevation above normal range)
   * Thrombocytopenia with platelet count < 50x10e9/L or more than 50% decrease in platelet count from the highest value achieved after transplant
   * Anemia below lower limit of normal or anemia requiring transfusion support as per center standard
   * Schistocytes on peripheral blood smear (>2 per HPF) OR histologic evidence of microangiopathy
   * Absence of coagulopathy (no uncompensated disseminated intravascular coagulation, DIC) at screening
5. The presence of TAM high risk features at baseline (or screening if baseline visit is skipped): Patients ≤ 16 years must have a Lansky score of ≤ 70 and patients > 16 must have Karnofsky score ≤ 70% and/or proteinuria (> 30 mg/dL) measured in two urine spot analyses.
6. Hypertension, defined for adults by SBP ≥ 160 mmHg and/or DBP ≥ 100 mmHg at baseline (or screening if baseline visit is skipped), and for pediatric patients by blood pressure greater than the 95th percentile for age, sex, and height (see Table 16-1). Additionally, patients who were started on antihypertensive medication after HSCT or who have received additional antihypertensive medication after HSCT will be eligible, even if they don't have elevated blood pressure.
7. Able to receive antibiotic prophylaxis against N. meningitides for the duration of the study.
8. Meningococcal vaccine(s) prior to LFG316 treatment if prior vaccination cannot be confirmed. The choice of vaccine(s) should take into account the serotypes prevalent in the geographic areas in which study patients will be enrolled. In case vaccination is not possible or will result in an unfavorable risk benefit ratio as judged by the investigator, vaccination can be postponed until deemed likely to be effective.
9. Patients <18 years old should receive vaccination for the prevention of S. pneumoniae and H. influenzae type b prior to LFG316 administration. In case vaccination is not possible or will result in an unfavorable risk benefit ratio as judged by the investigator, vaccination can be postponed until deemed likely to be effective.
10. Weight of at least 10kg.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or until the expected PD effect has returned to baseline, whichever is longer; or even longer if required by local regulations. Concomitant investigational treatment, including treatment in the context of a clinical trial with marketed drugs (off-label) may be acceptable but requires approval by the sponsor on the case by case basis.
2. Known hypersensitivity to any constituent of the study medication.
3. Patients with steroid refractory graft versus host disease (SRGvHD). SRGvHD is defined as progression (=increase in overall grade) after 5 days on ≥2mg/kg methylprednisolone or equivalent OR no improvement (no decrease in overall grade) after 10 days on ≥ 2mg/kg methylprednisolone or equivalent. If patients are receiving steroids for GvHD prophylaxis as per center standard, progression after 5 days and no response after 10 days after doubling the steroid dose will be regarded as steroid refractory.
4. Patients with ALT > 10x ULN at screening.
5. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (at screening or baseline).
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 45 days after stopping study medication. Highly effective contraception methods include:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (i.e., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
   * Female sterilization (have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization (at least 6 m prior to screening). The vasectomized male partner should be the sole partner for that subject.
   * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
   * In case of use of oral contraception women should have been stabile on the same pill for a minimum of 3 months before taking study treatment.
7. Sexually active males unwilling to use a condom during intercourse while taking drug and for 45 days after stopping investigational medication. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid. Male patients should not father a child in this period.
8. Positive HIV (ELISA and Western blot) test result (checked at screening). Historical local data will be acceptable if it the test was done within one month before start of HSCT conditioning and not more than 3 months before study visit 3.
9. A positive Hepatitis B surface antigen or Hepatitis C test result at screening. Historical local data will be acceptable if it the test was done within one month before start of HSCT conditioning and not more than 3 months before study visit 3.
10. Patients with any severe, progressive or uncontrolled acute or chronic medical condition (such as uncontrolled infectious disease or sepsis) or clinical laboratory abnormalities that in the investigator's opinion would make the patient inappropriate for entry into this study (at screening or baseline).
11. Patients with proven TTP as per historical data (as defined by ADAMST13 activity test) and if already available results of ADAMST13 test done at screening.
12. Patients previously treated with eculizumab for TAM.
13. Patients with known or suspected hereditary complement pathway deficiency. This exclusion criterion is not applicable to patients with complement pathway abnormalities/upregulation known to be associated with increased risk of transplant associated microangiopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Bucher, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (2):
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
- France (2):
  - Novartis Investigative Site, Paris, Cedex 10
  - Novartis Investigative Site, Marseille
- Germany (2):
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to low confidence of clinical benefit, this study was closed. In the beginning 3 participants were assigned to LFG316 on top of SoC & 4 subjects to only SoC (so total 7 randomized). 2 were randomized to SoC switched arm to LFG316 plus SoC. This means that 2 SoC and 2 in SoC then LFG316 are the same subjects as All SOC first.
Groups:
- LFG316 Plus Standard of Care (SoC): LFG316 plus SoC (excluding plasmapheresis and prohibited treatment)
Period: Overall Study
Arm/Group | LFG316 Plus Standard of Care (SoC) | All SoC First
Started | 3 | 4
Completed | 0 | 2
Not Completed | 3 | 2
Not completed — Patient/guardian decision | 1 | 0
Not completed — Death | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LFG316 Plus Standard of Care (SoC) | All SoC First | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.50) | 43.3 (8.54) | 49.4 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Schistocytes Per 1,000 Red Blood Cells (RBCs) for Hematological Responder Rate at 17 Weeks
Description: Hematological response rate was to be assessed at 17 weeks. However, due to early termination and with too few patients for statistical inference, the comparison between the two treatment arms LFG316 and SoC was not performed, and only descriptive statistics at different visits are provided for schistocytes Schistocytes <2/microscopic high power field (HPF) showed a hematological response
Time Frame: 17 weeks
Population: Only seven adult patients were enrolled prior to the early study termination decision. Due to low confidence of clinical benefit, this study was closed. There was too few patients for statistical inference.
Measure: Mean (Standard Deviation); unit: Number of Schistocytes per 1,000 RBCs
Arm/Group | LFG316 Plus Standard of Care (SoC) | All SoC First
Number analyzed (Participants) | 3 | 4
Number of Schistocytes per 1,000 RBCs
  Baseline (Day1) | 3.33 (2.082) | 7.25 (4.193)
  Day 2 | 4.33 (3.055) | 7.75 (7.042)
  Day 5 | 8.33 (6.506) | 7.25 (8.770)
  Day 8: number analyzed (Participants) | 3 | 3
  Day 8 | 12.67 (10.970) | 5.00 (1.732)
  Day 9: number analyzed (Participants) | 3 | 3
  Day 9 | 4.33 (4.933) | 8.33 (2.082)
  Day 12 | 7.00 (2.646) | 6.75 (7.676)
  Day 15 | 8.67 (11.590) | 6.00 (4.967)
  Day 16: number analyzed (Participants) | 3 | 3
  Day 16 | 7.33 (10.116) | 4.00 (1.00)
  Day 19: number analyzed (Participants) | 3 | 2
  Day 19 | 4.17 (5.107) | 9.50 (4.95)
  Day 29: number analyzed (Participants) | 3 | 2
  Day 29 | 12.00 (13.000) | 3.50 (2.121)
  Day 36: number analyzed (Participants) | 3 | 2
  Day 36 | 3.67 (1.528) | 4.00 (4.243)
  Day 43: number analyzed (Participants) | 3 | 1
  Day 43 | 8.67 (5.33) | 2.00
  Day 50: number analyzed (Participants) | 3 | 2
  Day 50 | 5.00 (3.464) | 5.00 (5.657)
  Day 57: number analyzed (Participants) | 3 | 1
  Day 57 | 19.00 (21.166) | 1.00
  Day 64: number analyzed (Participants) | 3 | 2
  Day 64 | 8.83 (8.780) | 10.50 (12.021)
  Day 71: number analyzed (Participants) | 1 | 2
  Day 71 | 2.00 | 12.00 (14.142)
  Day 78: number analyzed (Participants) | 1 | 2
  Day 78 | 2.00 | 14.50 (16.263)
  Day 85: number analyzed (Participants) | 0 | 2
  Day 85 |  | 4.00 (4.243)
  Day 92: number analyzed (Participants) | 0 | 2
  Day 92 |  | 2.50 (0.707)
  Day 99: number analyzed (Participants) | 0 | 1
  Day 99 |  | 4.00
  Day 106: number analyzed (Participants) | 0 | 2
  Day 106 |  | 3.50 (3.536)

2. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Peak plasma concentration (Cmax) Only seven adult patients were enrolled prior to the early study termination decision. Due to low confidence of clinical benefit, this study was closed. There was too few patients for statistical inference therefore only summary statistics of serum PK values at Day 1 and not at 52 Weeks
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LFG316 Plus Standard of Care (SoC) | All SoC First
Number analyzed (Participants) | 3 | 4
ng/mL | 440 (177) | 316 (53.7)

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC Last)
Description: Area under the plasma concentration versus time curve (AUC last) AUC up to the last measurable concentration. Only seven adult patients were enrolled prior to the early study termination decision. Due to low confidence of clinical benefit, this study was closed. There was too few patients for statistical inference therefore only summary statistics of serum PK values at Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | LFG316 Plus Standard of Care (SoC) | All SoC First
Number analyzed (Participants) | 3 | 4
h*μg/mL | 48400 (15000) | 19200 (21200)

4. Secondary Outcome: Time to Reach the Maximal Concentration (Tmax)
Description: Time to reach the maximal concentration (Tmax)Only seven adult patients were enrolled prior to the early study termination decision. Due to low confidence of clinical benefit, this study was closed. There was too few patients for statistical inference therefore only summary statistics of serum PK values at Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | LFG316 Plus Standard of Care (SoC) | All SoC First
Number analyzed (Participants) | 3 | 4
hours | 2.73 [2.18 to 2.92] | 2.67 [2.25 to 3.08]

5. Secondary Outcome: Complete Response Rate at 17 Weeks
Description: Complete response rate was planned to be assessed at 17 weeks. However, due to early termination and low sample size the comparison between the two treatment arms LFG316 and SoC was not performed. Only seven adult patients were enrolled prior to the early study termination decision. Due to low confidence of clinical benefit, this study was closed. There was too few patients for statistical inference.
Time Frame: 17 weeks
Population: Only 7 adult patients were enrolled prior to the early study termination. Due to low confidence of clinical benefit, this study was closed. There was too few patients for statistical inference and no data was reported.
Arm/Group | LFG316 Plus Standard of Care (SoC) | All SoC First
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Non-relapse Mortality
Description: Time to non-relapse-related mortality up to 17 weeks was not assessed due to the paucity of data. Only seven adult patients were enrolled prior to the early study termination decision. Due to low confidence of clinical benefit, this study was closed. There was too few patients for statistical inference.
Time Frame: 52 weeks
Population: as for outcome 5
Arm/Group | LFG316 Plus Standard of Care (SoC) | All SoC First
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) 21-April-2016 until Last Patient Last Visit (LPLV) 30-June-2017. All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to 1 year.
Description: Three patients died during the study. One patient from the LFG316 only group died due to sepsis that was considered related to the study drug per Investigator assessment. Two patients who switched from SoC to LFG316 died 5 and 9 days after switching, one due to respiratory failure and one due to thrombotic microangiopathy. However,for one patient the reason for discontinuation was reported as AE instead of death.
Groups:
- Standard of Care SoC: Standard of Care (SoC)
- SoC Then LFG316: SoC then LFG316
Arm/Group | LFG316 Plus Standard of Care (SoC) | Standard of Care SoC | SoC Then LFG316 | All SoC First
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/2 | 1/2 | 1/4
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/2 | 2/2 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LFG316 Plus Standard of Care (SoC) (N=3) | Standard of Care SoC (N=2) | SoC Then LFG316 (N=2) | All SoC First (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 1 | 0 | 1
Graft versus host disease in liver (Immune system disorders) | 0 | 1 | 0 | 1
Graft versus host disease in skin (Immune system disorders) | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Microangiopathy (Vascular disorders) | 1 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LFG316 Plus Standard of Care (SoC) (N=3) | Standard of Care SoC (N=2) | SoC Then LFG316 (N=2) | All SoC First (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 1
Keratitis (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 2 | 1 | 3
Localised oedema (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 2 | 2 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Graft versus host disease in skin (Immune system disorders) | 0 | 1 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 2 | 0 | 2
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 1
Pertussis (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 2
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 1 | 1 | 2
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 1
Norovirus test positive (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1
Psychotic behaviour (Psychiatric disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Anuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 2 | 0 | 1 | 1
Hypotension (Vascular disorders) | 2 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 2 | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02763644/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT02763644/SAP_001.pdf